CLINICAL TRIAL: NCT03592706
Title: A Phase II/III Clinical Trial With Ex Vivo Expanded Autologous Immune Killer Cells to Treat Liver Cancer Patients as an Adjunct Therapy
Brief Title: Autologous Immune Killer Cells to Treat Liver Cancer Patients as an Adjunct Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ivy Life Sciences, Co., Ltd (Industry)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVY02; NCT01024530 (obsolete NCT alias)
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: HepatoCellular Carcinoma; Liver Cancer
Keywords: HepatoCellular Carcinoma; Liver Cancer; Immune Killer Cells; IKC; Immune Therapy; Immunotherapy; Cell Therapy; IVY; IVY02
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IKC and TACE (Experimental): IKC (Immune Killer Cells) and TACE(Transcatheter Arterial Chemoembolization)
  Interventions: Biological: IKC (Immune Killer Cells); Procedure: TACE (Transcatheter Arterial Chemoembolization)
- TACE (Active Comparator): TACE (Transcatheter Arterial Chemoembolization)
  Interventions: Procedure: TACE (Transcatheter Arterial Chemoembolization)

INTERVENTIONS:
Biological: IKC (Immune Killer Cells)
  Other Names: Autologous Immune Killer Cells
  Arms: IKC and TACE
Procedure: TACE (Transcatheter Arterial Chemoembolization)
  Other Names: TACE

SUMMARY:
The purpose of this study is to evaluate the efficacy of ex vivo expanded autologous immune killer cells in treating hepatocellular carcinoma patients in：

1. Reduction of tumor size
2. Reducing the relapse rate: Reducing the frequency of TACE treatment by IKC injections.

DETAILED DESCRIPTION:
This is a phase II/III clinical study. Blood is drawn from the patient and brought to our laboratory for isolation of immune cells. These immune cells are then proliferated over a two week period and used to produce the patented product IKC (Immune Killer Cells). The IKC will then infused back into the patient to treat the cancer. Each patient will receive a total of twelve infusions.

60 patients are anticipated to be recruited. This is a double-arm study, the experimental group will receive IKC treatment along with TACE treatment. The control group will receive only TACE treatment. 30 patients will be randomized into each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Sign and give written informed consent.
2. Age≧20 years, but<80 years.
3. Hepatocellular carcinoma by CT, MRI, AFP, angiography or cytology/biopsy examinations.
4. Barcelona staging system stage B and C.
5. Never receive TACE treatment and comply with the standard of TACE treatment.
6. Child-Pugh stage A and B.
7. ECOG performance status 0 to 2.

Exclusion Criteria:

1. Participant of other clinical trial within the past 4 weeks of screening period.
2. Receiver of chemotherapy, radiotherapy, immunotherapy, hormone therapy, local tumor therapy, or target therapy within the past 4 weeks of screening period.
3. Carriers of HIV or HTLV within the past 4 weeks of screening period.
4. With Active acute or chronic infection by (investigator's judgement).
5. Other diseases, except hepatocellular carcinoma, which are life-threatening to the patients (by investigator's judgement) for example:

   5.1 Active cardiac disease requiring therapy for coronary artery disease, congestive heart failure, arrhythmia or myocardial infarction.

   5.2 With previous history of encephalopathy within the past six months.

   5.3 Involved Involving systemically or known central nerve system diseases(brain or meningeal metastasis).
6. Women of pregnant or breast-feeding or child-bearing potential but without adequate contraception.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-12 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change of tumor size | One year
  Evaluate the efficacy of autologous immune killer cells using Response Evaluation Criteria in Solid Tumors (RECIST) by recording net changes of tumor sizes
Progression-Free Survival (PFS) | One year
  The length of time during and after the treatment of a disease, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Improvement of immune responses | One year
  Evaluate the efficacy and safety of in vitro proliferating autoimmune killer cells as adjuvant therapy for the treatment of liver cancer patients and promote anti-cancer immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Bao Hsieh, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri Service General Hospital, Taipei, Taiwan